CLINICAL TRIAL: NCT03534102
Title: Can Simplified and More Detailed Instructions Affect Post-Operative Narcotic Consumption
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to limitations caused by COVID, enrollment targets could not be met.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Wolfgang Fitz, M.D., Associate Orthopedic Surgeon, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OpioidTaperingTKR/THR
Record Dates: First submitted 2018-04-24; First posted 2018-05-23 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Opioid Use; Opioid Dependence; Knee Pain Chronic; Knee Osteoarthritis
Keywords: Total Hip Arthroplasty; Total Knee Arthroplasty; Opioid Dependence; Opioid Tapering
MeSH Terms: conditions — Opioid-Related Disorders; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Testing 3 sequential standards of care; each of 3 arms lasts 4 months, and all patients recruited within an arm are assigned to the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard of Care (No Intervention): Standard instructions from hospital. Subjects talk with hospital staff only when they call the hospital, when RA calls at various benchmarks, and at postoperative clinic visits. Subjects record opioid tapering in diary.
- Improved Instructions (Experimental): Improved opioid-tapering instructions given upon discharge from hospital. Subjects talk with hospital staff only when they call the hospital, when RA calls at various benchmarks, and at postoperative clinic visits. Subjects record opioid tapering in diary.
  Interventions: Drug: Improved Opioid-Tapering Instructions
- Improved Instructions and Educator (Experimental): Improved opioid-tapering instructions given upon discharge from hospital. Subject receives regular phone calls from educator for counseling in opioid tapering. Subjects record opioid tapering in diary.
  Interventions: Drug: Improved Opioid-Tapering Instructions; Behavioral: Clinical Patient Educator

INTERVENTIONS:
Drug: Improved Opioid-Tapering Instructions — Applied to first and second experimental groups in the form of discharge instructions and directions from nursing staff.
  Arms: Improved Instructions; Improved Instructions and Educator
Behavioral: Clinical Patient Educator — Applied to second experimental group in the form of regular calls about weaning off narcotic medications.
  Arms: Improved Instructions and Educator

SUMMARY:
This project intends to investigate whether (1) a patient-maintained opioid diary provides an accurate measure of opioid consumption (morphine equivalents), (2) improved patient educational materials decrease narcotic consumption, and (3) using a pain management counselor provides additional benefits in decreasing narcotic consumption when used in conjunction with improved educational materials. Furthermore, the investigators would like to investigate the effect of the patient-maintained diaries, the improved educational materials, and the pain management counselor on pain levels, nausea, sleep quality, and patient satisfaction.

All patients undergoing orthopedic surgery at Brigham and Women's Faulkner Hospital and choose to participate will be assigned to a treatment group based on which arm of the study is being tested at the time; (the treatment arms are sequential). Members of Group 1 (control group) will receive the current standardized institutional discharge care for orthopedic surgery and an added tracking diary. Members of Group 2 (experimental group 1) will receive more detailed educational materials regarding postoperative pain management - including instructions to how to taper their narcotic usage - as well as a tracking diary. Members of Group 3 (experimental group 2) will receive not only the educational materials of Group 2, but also weekly phone calls from a clinical patient educator to remind them of proper use of the diary and narcotic tapering.

DETAILED DESCRIPTION:
This project intends to investigate whether (1) a patient-maintained opioid diary provides an accurate measure of opioid consumption (morphine equivalents), (2) improved patient educational materials decrease narcotic consumption, and (3) using a pain management counselor provides additional benefits in decreasing narcotic consumption when used in conjunction with improved educational materials. Furthermore, the investigators would like to investigate the effect of the patient-maintained diaries, the improved educational materials, and the pain management counselor on pain levels, nausea, sleep quality, and patient satisfaction. The enrollment of the study will depend on the amount of patients that fall into each treatment arm - each of which will last for a fixed period of time. The expected enrollment is approximately 1000-1200 patients.

All patients undergoing orthopedic surgery at Brigham and Women's Faulkner Hospital and meet all eligibility criteria will be informed about the study and asked whether they would like to participate. Those who agree will be assigned to a treatment group based on which arm of the study is being tested at the time (the treatment arms are sequential). Members of Group 1 (control group) will receive the current standardized institutional discharge care for orthopedic surgery and an added tracking diary. Members of Group 2 (experimental group 1) will receive more detailed educational materials regarding postoperative pain management - including instructions to how to taper their narcotic usage - as well as a tracking diary. Members of Group 3 (experimental group 2) will receive not only the educational materials of Group 2, but also regular phone calls from a clinical patient educator to remind them of proper use of the diary and narcotic tapering.

Each enrolled patient will be given verbal and written (printed and/or electronic format) instructions about narcotic medication by the nursing staff upon hospital discharge. The instructions will explain when to use such medications, how to taper off them, and how to document them. Following discharge, patients will record their opioid consumption on their own and document their pain, nausea, sleep and satisfaction. At the first post-operative appointment, patients' levels of opioid use will be recorded and actual tablets consumed compared with prescription received. If they receive a new prescription they will receive a matching diary for the total length of planned opioid treatment, including directions on how to wean themselves off the opioids. Outcome measures will be collected at both post-operative visits, the first a week after surgery and the second 2-3 months following. Additional data including length of stay, postoperative complications including infection and readmission, Emergency Department visits, and routinely collected postoperative functional outcome measures (PROMs) will be recorded.

The Principal Investigator (PI) will review all pain, satisfaction, narcotic usage and proprioception data on a weekly basis with the research assistant (RA) as it is collected. These checks will help to ensure validity and patient safety. Privacy and confidentially will be assured by using codes as deidentifiers in place of identifying information on any data sheets used in analysis. Data which identifies the patient will be made available only to investigators and stored only in a private folder on department computers protected with a firewall. No data will be shared outside of Partners. Adverse events will be promptly reported to the Partners Human Research Committee (PHRC) as per PHRC rules.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Date of surgery between 3 weeks and 8 weeks away
* Undergoing total hip or total knee replacement [including simultaneous bilateral]
* Eligible based on our standard Faulkner Hospital pre-op assessment

Exclusion Criteria:

* If female, pregnant
* Undergoing partial joint replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-06 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption: Amount | 2-3 months following surgery, or as needed (total usage assessed after postoperative appointments).
  Total amount of patients' opioid consumption, measured in mg of morphine equivalents.
Opioid Usage After One Week | 7 days following surgery.
  The proportion of patients who have finished taking opioids by the first postoperative appointment, approximately one week after surgery.
Total Opioid Consumption: Days | 2-3 months following surgery, or as needed (total usage assessed after postoperative appointments).
  The total number of days in which each patient took opioid medications after surgery.

SECONDARY OUTCOMES:
Opioid Usage After Two Weeks | 14 days following surgery.
  The proportion of patients who have finished taking opioids two weeks after surgery.
Visual Analogue Scale (VAS) Score 1: "How much pain do you feel in your operative site when resting?" | 2-3 months following surgery (measured at second postoperative appointment).
  Surgical site pain. Scale 0-10, with 0 best and 10 worst.
VAS Score 2: "How much pain do you feel in your operative site when moving?" | 2-3 months following surgery (measured at second postoperative appointment).
  Surgical site pain. Scale 0-10, with 0 best and 10 worst.
VAS Score 3: "How well are you sleeping?" | 2-3 months following surgery (measured at second postoperative appointment).
  Sleep quality. Scale 0-10 with 0 worst and 10 best.
VAS Score 4: "How bad is your nausea?" | 2-3 months following surgery (measured at second postoperative appointment).
  Nausea. Scale 0-10, with 0 best and 10 worst.
VAS Score 5: "How satisfied are you with your pain management?" | 2-3 months following surgery (measured at second postoperative appointment).
  Satisfaction. Scale 0-10 with 0 worst and 10 best.
Questionnaire Answers | 3 months after surgery.
  Questionnaire given to patients 3 months after surgery. Patients are asked about how opioid medications are typically stored and consumed at home.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fitz, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Faulkner Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon DB, de Leon-Casasola OA, Wu CL, Sluka KA, Brennan TJ, Chou R. Research Gaps in Practice Guidelines for Acute Postoperative Pain Management in Adults: Findings From a Review of the Evidence for an American Pain Society Clinical Practice Guideline. J Pain. 2016 Feb;17(2):158-66. doi: 10.1016/j.jpain.2015.10.023. Epub 2015 Dec 21. PMID 26719073
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Reynolds MA. Postoperative pain management discharge teaching in a rural population. Pain Manag Nurs. 2009 Jun;10(2):76-84. doi: 10.1016/j.pmn.2008.07.003. Epub 2009 Jan 4. PMID 19481046
- [Background] Wakim JH. Alleviating symptoms of withdrawal from an opioid. Pain Ther. 2012 Dec;1(1):4. doi: 10.1007/s40122-012-0004-5. Epub 2012 Sep 20. PMID 25134933
- [Background] Ninkovic J, Roy S. Morphine decreases bacterial phagocytosis by inhibiting actin polymerization through cAMP-, Rac-1-, and p38 MAPK-dependent mechanisms. Am J Pathol. 2012 Mar;180(3):1068-1079. doi: 10.1016/j.ajpath.2011.11.034. Epub 2012 Jan 14. PMID 22248582
- [Background] Goesling J, Moser SE, Zaidi B, Hassett AL, Hilliard P, Hallstrom B, Clauw DJ, Brummett CM. Trends and predictors of opioid use after total knee and total hip arthroplasty. Pain. 2016 Jun;157(6):1259-1265. doi: 10.1097/j.pain.0000000000000516. PMID 26871536
- See also: Carr DB, Morlion B. Pain After Surgery: What Health-Care Professionals Should Know. — https://www.europeanpainfederation.eu/wp-content/uploads/2017/01/02.-What-Health-Care-Professionals-Should-Know-About-Pain-After-Surgery.pdf